CLINICAL TRIAL: NCT01282749
Title: The Hospitals-Churches Partnership for Health Project: SisterTalk Hartford
Brief Title: Effectiveness of SisterTalk Hartford for Weight Loss Among African-American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: St. Francis Hospital & Medical Center, Hartford CT (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: O02-07-003-E; SR0550 (Other: Saint Francis Hospital)
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; African American; Women; Translational; Faith based; Community based participatory research
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SisterTalk Hartford First (Experimental): 12-week group support and film-based healthy lifestyle education program, including information on healthy nutrition and food preparation, increasing activity and exercise, healthy lifestyle behavior modification, and supportive spiritual materials.
  Interventions: Behavioral: SisterTalk Hartford
- SisterTalk Hartford Second (Other): Participants received general film series on healthy lifestyles while waiting to participate in the experimental arm.
  Interventions: Behavioral: Attention control video series

INTERVENTIONS:
Behavioral: SisterTalk Hartford — 12-week group support and film-based healthy lifestyle education program, including information on healthy nutrition and food preparation, increasing activity and exercise, healthy lifestyle behavior modification, and supportive spiritual materials.
  Arms: SisterTalk Hartford First
Behavioral: Attention control video series — Participants received general film series on healthy lifestyles while waiting to participate in the experimental arm.
  Arms: SisterTalk Hartford Second

SUMMARY:
The purpose of the SisterTalk Hartford study was to assess whether a theoretically- and scientifically-based, culturally acceptable weight loss program could be effectively translated into a faith-based program and subsequently delivered in the church to help African-American women lose weight.

ELIGIBILITY:
Inclusion Criteria:

* BMI of at least 25.0
* self-identifies as Black or African-American
* able to do mild physical activity such as walking or chair exercises

Exclusion Criteria:

* has insulin dependent diabetes
* is pregnant, nursing, or had a baby in the past 4 months
* has ever been treated for an eating disorder (e.g. anorexia nervosa, bulimia)
* had a heart attack in the past 2 years requiring hospitalization
* has ever had a stroke
* has congestive heart failure
* has uncontrolled hypertension
* currently participating in another study
* is on a doctor-prescribed diet that cannot be changed (e.g. very low protein diet for a person in liver failure)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2002-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
weight loss | assessed 4 times over 2 years, in roughly 6 mo intervals
  Change in BMI

CONTACTS AND LOCATIONS:
Overall Officials: Judith Fifield, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States